# **Informed Consent Form**

Amasya University, Faculty of Medicine Sabuncuoğlu Şerefeddin Training and Research Hospital

#### **Study Title:**

Effect of Dexmedetomidine on Recurrent Laryngeal Nerve Monitoring: A Comparative Study With Midazolam

#### **Principal Investigator:**

Dr. Suat Evirgen, Department of General Surgery Amasya University, Faculty of Medicine

### **Purpose of the Study**

You are being invited to participate in this research study because you are scheduled for thyroid surgery. The purpose of this study is to compare the effects of two commonly used anesthetic agents, dexmedetomidine and midazolam, on monitoring the recurrent laryngeal nerve during surgery. This monitoring helps the surgeon identify and protect the nerves controlling your vocal cords.

#### **Procedures**

If you agree to participate, you will undergo thyroid surgery under general anesthesia as already planned. During anesthesia, you will receive either dexmedetomidine or midazolam, in addition to standard medications. Throughout the surgery, special monitoring will be used to record nerve signals. Data on nerve monitoring, heart rate, blood pressure, recovery, and possible side effects will be collected. No additional invasive procedures will be performed other than what is normally required for your operation.

#### **Risks and Discomforts**

Both dexmedetomidine and midazolam are standard anesthetic medications. Possible risks include changes in heart rate, blood pressure, drowsiness, or delayed recovery. These are routinely managed in the operating room. There are no additional risks beyond standard thyroid surgery and anesthesia.

#### **Benefits**

There may be no direct benefit to you. However, the information gained may help improve anesthesia protocols and enhance patient safety in future thyroid surgeries.

# **Confidentiality**

Your personal information will remain confidential. Data collected will be coded and analyzed without identifying you by name. Only the research team will have access to your records. Results may be published in medical journals, but your identity will never be revealed.

## **Voluntary Participation**

Your participation in this study is entirely voluntary. You may refuse to participate or withdraw at any time without affecting your medical care or your relationship with your doctors.

## **Contacts for Questions**

If you have questions about the study, please contact:

**Dr. Suat Evirgen** – Department of General Surgery, Amasya University

Phone: +90 (532) 551 8900 Email: opdrse@gmail.com

If you have questions about your rights as a participant, you may contact the Amasya University Non-Interventional Clinical Research Ethics Committee.